CLINICAL TRIAL: NCT02018445
Title: Accell Evo3™ Demineralized Bone Matrix in Instrumented Lumbar Spine Fusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SeaSpine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ACC3-US-2012-2
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Results first posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Degenerative Changes; Stenosis; Spondylosis
MeSH Terms: conditions — Constriction, Pathologic; Spondylosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Accell Evo3 DBM & Local Autograft (Other): Accell Evo3 DBM (posterolateral gutter symptomatic side) and Local Autograft (posterolateral gutter contralateral non-symptomatic side)
  Interventions: Procedure: Posterolateral Fusion

INTERVENTIONS:
Procedure: Posterolateral Fusion

SUMMARY:
The objective of this study is to prospectively evaluate the performance of Integra Accell Evo3 Demineralized Bone Matrix as an adjunct for instrumented posterolateral spine fusion, as compared to local autograft.

ELIGIBILITY:
Inclusion Criteria:

1. Are 18 (eighteen) years of age or older at the time of surgery.
2. Require spinal fusion using Transforaminal Lumbar Interbody Fusion (TLIF), Posterior Lumbar Fusion (PLF) or Posterior Lumbar Interbody Fusion (PLIF), with or without the use of an interbody spacer, at 1 to 3 levels between L3-S1.
3. Willing and able to return for the scheduled follow-up visits, follow post-operative instructions and undergo the required radiographic exams (A/P, Lateral Neutral and Lateral Flexion/Extension X-rays) for up to 4 time points between 2 weeks and 12 months post-surgery (3 months ± 2 weeks, 6±1 months, 12±2 months and if required 24±3 months post-surgery), including one CT-scan at 12±2 months.
4. Unresponsive to conservative care over a period of at least 6 months or has signs and/or symptoms that mandate urgent surgical intervention.
5. Willing and able to sign study specific informed consent.

Exclusion Criteria:

1. Are long term users of medications (i.e. steroids greater than 8 days) that are known to inhibit fusion or bone metabolism at any time within 6 months prior to surgery. Exceptions are inhaled steroids for asthma treatment (i.e. subjects on inhaled steroids are allowed), or epidural steroid injections.
2. Are taking immunosuppressive agents (Cancer chemotherapy, treatment with Disease Modifying Anti-rheumatic drugs (DMARDs) or any similar immunomodulating drugs) or are treated with Growth Factors or Insulin at any time within 6 months prior to surgery.
3. Are being treated with radiotherapy.
4. Are having medical conditions, known to impact bone metabolism, such as Paget's disease, osteoporosis, severe degenerative bone disease.
5. Are smokers and/or nicotine/tobacco users.
6. Have a Body Mass Index (BMI) ≥ 40
7. Are pregnant, lactating or women wishing to become pregnant.
8. Are a prisoner.
9. Are currently participating in an investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the study endpoints.
10. Prior spine surgery at the index level except posterior decompressive surgery where the posterior elements are preserved e.g. facet saving techniques such as discectomy, laminotomy, and intradiscal procedures.
11. Use of any other bone graft or bone graft substitute in addition to or in place of Accell Evo3 and/or local autograft.
12. Use of routine prophylactic NSAIDS for 3 months post-operatively, but low dose concomitant pain medications e.g. aspirin should be continued and recorded on the Concomitant Pain Medications case report form (CRF).
13. Have a known sensitivity Polymyxin Sulfate B, Bacitracin, Gentamycin and/or Iodine.
14. Severe vascular or neurological disease.
15. Uncontrolled diabetes.
16. Uncooperative patients who will not or cannot follow postoperative instructions, including individuals who abuse drugs and/or alcohol.
17. Renal impairment.
18. Active or latent infection in or around the surgical site.
19. Accell Evo3 is contraindicated when there is significant vascular impairment proximal to the implantation site and when there are metabolic or systemic bone disorders that affect bone or wound healing, or when stabilization of the defect is not possible.
20. The use of Accell Evo3 is also contraindicated in cases where intraoperative soft tissue coverage is not planned or possible and in infected or contaminated wounds.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-11; Primary Completion 2015-07 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Yuan, M.D, Principal Investigator — Memorial Orthopaedic Surgical Group
Locations (1):
- Memorial Orthopaedic Surgical Group, Long Beach, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the study in which each patient undergoes posterolateral fusion (PLF). During PLF, each spinal level is treated with two graft materials, the symptomatic posterolateral gutter is treated with study arm (Accel Evo3) and the contralateral non-symptomtic posterolateral gutter is treated with the control arm (local autograft).
Groups:
- All Patients: Posterolateral fusion study in which each patient undergoes posterolateral fusion (PLF). During the PLF, each spinal level is treated with two graft materials, the symptomatic posterolateral gutter is treated with study arm (Evo3) and the contralateral posterolateral gutter is treated with the control arm (local autograft).
Period: Overall Study
Arm/Group | All Patients
Started | 36
Completed | 29
Not Completed | 7

BASELINE CHARACTERISTICS:
Units Other Than Participants: Spinal Levels
Arm/Group | All Patients
Number analyzed (Participants) | 29
Number analyzed (Spinal Levels) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 9
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.39 (5.38)

OUTCOME MEASURES:

1. Primary Outcome: Time to Arthrodesis (Fusion) for Each Spinal Level (Unit), as Measured by X-rays.
Description: There were 29 patients and 43 total spinal levels (unit) treated at baseline. Time to arthodesis was measured as the mean time to achieve fusion. At each time point fusion was evaluated, the first time point fusion was achieved was considered fusion.
Time Frame: 12 months
Population: Time to arthodesis was measured as the mean time to achieve fusion for each spinal level treated.
Measure: Mean (Standard Deviation); unit: months to fusion
Units Other Than Participants: Spinal Levels
Groups:
- All Patients: Posterolateral fusion: each spinal level is treated with two graft materials, the posterolateral gutter is treated with study arm (Accel Evo3) and the contralateral posterolateral gutter is treated with the control arm (local autograft).
Arm/Group | All Patients
Number analyzed (Participants) | 29
Number analyzed (Spinal Levels) | 43
months to fusion | 6 (5.7)

2. Secondary Outcome: Percent (%) of Fusion for Each Spinal Level (Unit), as Measured by Computed Tomography (CT) Scan
Time Frame: 12 months
Measure: Count of Units; unit: Posterolateral Sides
Units Other Than Participants: Posterolateral Sides
Arm/Group | All Patients
Number analyzed (Participants) | 34
Number analyzed (Posterolateral Sides) | 34
Posterolateral Sides | 26

3. Secondary Outcome: Medical Outcomes: Oswestry Disability Index (ODI)
Description: The ODI is an index derived from the Oswestry Low Back Pain Questionnaire used by surgeons, clinicians and researchers to quantify disability for low back pain. The questionnaire is self-completed and covers 10 topics about pain intensity, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Scores are from 0-100 and a lower score represents a better score.
Time Frame: 12 months
Population: Patients were lost to follow-up as study progressed
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- All Patients: Patients were treated at multiple levels. Accell Evo3 was placed in the posterolateral gutter of the symptomatic side and local autograft was used in the posterolateral gutter of the contralateral asymptomatic side.
Arm/Group | All Patients
Number analyzed (Participants) | 29
units on a scale
  Baseline | 47.6 (17.7)
  6 Month: number analyzed (Participants) | 27
  6 Month | 26.0 (16.9)
  12 Month: number analyzed (Participants) | 26
  12 Month | 25.0 (21.0)

4. Secondary Outcome: Medical Outcomes: Worst Leg Pain Visual Analog Scale (VAS)
Description: The visual analogue scale (VAS) is a commonly used outcome measure for research studies. It is presented as a 100-mm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "0"/no pain at all" and "100/worst pain imaginable." The study in this scale is used for the worst leg pain. A lower score represents a better score.
Time Frame: 12 months
Population: Patients lost to follow-up over course of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Patients
Number analyzed (Participants) | 29
units on a scale
  Baseline | 64.8 (28.8)
  6 Month: number analyzed (Participants) | 28
  6 Month | 15.3 (25.7)
  12 Month: number analyzed (Participants) | 26
  12 Month | 13.3 (25.2)

5. Secondary Outcome: Medical Outcomes: Back Pain Visual Analog Scale (VAS)
Description: The visual analogue scale (VAS) is a commonly used outcome measure for research studies. It is presented as a 100- mm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "0"/no pain at all" and "100/worst pain imaginable." The study in this scale is used for the back pain. A lower score represents a better score.
Time Frame: 12 months
Population: Patients were lost to follow-up as study progressed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Patients
Number analyzed (Participants) | 29
units on a scale
  Baseline Over Time: Baseline | 66.1 (30.6)
  6 Month: number analyzed (Participants) | 28
  6 Month | 23.6 (28.4)
  12 Month: number analyzed (Participants) | 26
  12 Month | 22.3 (30.2)

6. Secondary Outcome: Medical Outcomes: Measure of EQ-5D™ Visual Analog Scale (VAS).
Description: EQ-5D is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments. The EQ-5D consists of a descriptive system and the EQ VAS. The EQ-5D-5l has a descriptive system and the EQ visual analogue scale (EQ VAS). The EQ VAS records the patient's self-rated health on a vertical visual analogue scale. Only the EQ VAS Score was analyzed in the study. The EQ VAS scored from 0-100 and a lower score represents a better score.
Time Frame: 12 months
Population: Patients were loss to follow-up as clinical study progressed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Patients
Number analyzed (Participants) | 29
units on a scale
  Baseline | 73.0 (21.0)
  6 Month: number analyzed (Participants) | 28
  6 Month | 82.2 (13.5)
  12 Month: number analyzed (Participants) | 27
  12 Month | 81.8 (20.0)

7. Secondary Outcome: Medical Outcomes: Maintenance of Lower Extremity Neurological Function
Description: Posterolateral fusion study in which one spinal level is treated with both the study and control arm. One posterolateral spinal side is Evo3 and the other posterolateral spinal side is local autograft.
  NA (Not Applicable): Neurological function data was not able to be analyzed as there was a limitation of the method in the ability to distinguish between left and right side neurological function. Neurological function is indistinguishable between the right and left side of the lower extremities using the methods in the protocol and analysis of neurological function therefore would have made no impact on the outcome of the study.
Time Frame: 12 months
Population: NA (Not Applicable): Neurological function data was not able to be analyzed as there was a limitation of the method in the ability to distinguish between left and right side neurological function. Neurological function is indistinguishable between the right and left side of the lower extremities using the methods in the protocol.
Groups:
- All Patients: All patients
Arm/Group | All Patients
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Patients With Serious Adverse Events, Adverse Device Effects, Serious Adverse Device Effects and Subsequent Surgical Interventions
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 36
Participants | 8

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 8/36
Other Adverse Events (participants affected / at risk) | 17/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=36)
Infection (Infections and infestations) | 2 (2)
Fall resulting in injury (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain (Nervous system disorders) | 4 (5)
Alcohol Abuse (Social circumstances) | 1 (1)
Device (non-study) complication (Surgical and medical procedures) | 1 (1)
wound drainage (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=36)
Pain, stiffness, strain, or discomfort (Nervous system disorders) | 11 (13)
Minor fracture (Musculoskeletal and connective tissue disorders) | 2 (3)
Medication reaction (Immune system disorders) | 2 (2)
Device (non-study) Complication (Surgical and medical procedures) | 1 (1)
Minor cut (Skin and subcutaneous tissue disorders) | 2 (4)
Impacted bowel (Gastrointestinal disorders) | 1 (1)
Muscle tear (Musculoskeletal and connective tissue disorders) | 1 (1)
Fall on side with no reported outcome (Musculoskeletal and connective tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Radiographic Haloing of Screws (non-study) (Surgical and medical procedures) | 1 (1)
Left ear carcinoma removed (Skin and subcutaneous tissue disorders) | 1 (1)
Elevated blood pressure (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days